CLINICAL TRIAL: NCT01746628
Title: Intrauterine Use of FloSeal: Is it Safe and Useful?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David L Zisow MD LLC (Industry)
Responsible Party: Principal Investigator, David L Zisow, MD, Gynecologist and Assoc. Chief of Minimally Invasive Surgery, David L Zisow MD LLC
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1971
Record Dates: First submitted 2012-12-06; First posted 2012-12-11 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Operative Hemorrhage
Keywords: type 0 myomata; type 1 myomata; type 2 myomata; bleeding; hemorrhage; hysteroscopy; FloSeal
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage | interventions — Hysterectomy; FloSeal Matrix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hysterectomy without FloSeal (Placebo Comparator): Endometrial curettage Intrauterine foley balloon placement for 5 minutes Removal of intrauterine foley balloon Saline irrigation of uterine cavity Hysterectomy
  Interventions: Procedure: Hysterectomy with FloSeal
- Hysterectomy with FloSeal (Active Comparator): Endometrial curettage FloSeal placement into uterine cavity Intrauterine foley balloon placement for 5 minutes Removal of intrauterine foley balloon Saline irrigation of uterine cavity Hysterectomy
  Interventions: Procedure: Hysterectomy with FloSeal

INTERVENTIONS:
Procedure: Hysterectomy with FloSeal — Evaluation of the effects of intrauterine FloSeal
  Other Names: Endometrial curettage; FloSeal placement into uterine cavity; Intrauterine foley balloon placement for 5 minutes; Removal of intrauterine foley balloon; Saline irrigation of uterine cavity; Hysterectomy

SUMMARY:
When having certain types of outpatient surgery inside the uterine cavity some women experience heavy bleeding. The only method presently available for controlling such bleeding, short of removing the uterus, involves the placement of a balloon pressure device inside the uterine cavity. The pressure along with the patient's own natural clotting ability will generally stop the bleeding. However, this treatment usually requires at least a 24 hour stay in the hospital. The investigators are researching the use of a compound (FloSeal) already approved for use in other areas of the human body, as a method of controlling bleeding. The use of FloSeal in the uterine cavity has not yet been tested and therefore is not yet an FDA approved indication for its safe use to control bleeding from the uterine cavity. In this study, The investigators want to find out what effect(s) FloSeal has on the uterine cavity.

Twenty individuals will be included in this study at Northwest Hospital Center. All twenty individuals will be treated in the same fashion except ten of the participants will randomly be assigned to receive FloSeal and ten will not.

Study participants are individuals currently scheduled to have a hysterectomy procedure, which involves surgically removing the uterus from the body for a previously determined standard of care treatment for a non- cancerous medical problem. Before performing the hysterectomy and evaluating the effects of FloSeal upon the tissues within the uterine cavity the following will be done. Once under anesthesia the uterine cavity will be subjected to a curettage (sharp scrapping) to produce a minor amount of bleeding from the lining of the uterus. Ten of the 20 study participants, randomly chosen, will then have FloSeal placed into their uterine cavity. The study participants will not know whether they received FloSeal or not. A balloon pressure device will then be placed into the uterine cavity of all 20 individuals and left in place for 5 minutes. After the allotted time, the balloon device will be removed. The hysterectomy will then be completed appropriately using standard methods and techniques. The uterus, once removed will be evaluated pathologically to determine the effects of the FloSeal upon the tissues of the cavity in those so treated and compared to the same analysis in those individuals who did not receive FloSeal. The pathologist will not know which patients received or did not receive FloSeal.

This use of FloSeal is not currently an FDA approved use of the compound. The goal of this study is to obtain FDA approval for use in this situation.

DETAILED DESCRIPTION:
Patients will be followed until fully recovered from surgery, usually 6 to 8 weeks. Any complications will be duly noted and treated appropriately. The final end point for follow up will be when the patient is finally discharged from care having achieved what is usually perceived as a return to all normal activity.

ELIGIBILITY:
Inclusion Criteria:Women undergoing hysterectomy for non-malignant indications -

Exclusion Criteria:Malignancy Inability to remove uterus without morcellation

-

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Tissue effects of FloSeal upon endometrium on day 1 | Immediate post operative effects
  Pathological (microscopic and histochemical) evaluation of endometrial curettings and uterine specimens in all study cases to evaluate immediate (day 1) tissue effects of FloSeal upon the endometrium.

CONTACTS AND LOCATIONS:
Overall Officials: David L Zisow, MD, Principal Investigator — LifeBridge Health
Locations (1):
- Northwest Hospital, Randallstown, Maryland, United States